CLINICAL TRIAL: NCT06934369
Title: Development and Evaluation of a Multi-Component Intervention to Support HIV Care Engagement Among Patients Receiving Cancer Treatment in Zimbabwe
Brief Title: Improving Engagement in HIV and Cancer Care in Zimbabwe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michalina Montaño, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: RG1123169; K01MH132505 (NIH); NCI-2023-02951 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 11131 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Cancer; HIV
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a pre-post, quasi-experimental study design, consisting of an initial (pre-intervention) observational cohort, a period of intervention development and process improvement, and a second observational (post-intervention) cohort. The primary outcome of acceptability will be assessed only in the second cohort. Secondary outcomes will be compared between the pre-intervention and post-intervention cohorts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-intervention cohort (No Intervention): This is a pre-post study. The pre-intervention cohort will not experience any intervention. The barriers to HIV care experienced by the pre-intervention cohort will be documented and used to develop strategies to support engagement in HIV care during cancer treatment. After follow-up is complete for the pre-intervention cohort, we will implement the strategies to support engagement in HIV care at the Parirenyatwa Hospital Radiotherapy Centre.
- Post-intervention cohort (Experimental): The intervention will be developed based on barriers to HIV care experienced by the pre-intervention cohort. It will be a system intervention, implemented at the Radiotherapy Centre at Parirenyatwa Hospital. It may include strategies like improving documentation of HIV-related information in oncology patient records, improving processes for referrals and access to HIV-related prescriptions, and supporting better communication between oncology and HIV clinical care teams. These strategies will be implemented with a period of process improvement between the pre- and post-intervention cohorts. Because the intervention will change the health system, all new patients who begin cancer treatment after the intervention is implemented will experience the health system updates. We will begin enrollment in the post-intervention cohort after process improvement is complete.
  Interventions: Other: Strategies to improve HIV care engagement

INTERVENTIONS:
Other: Strategies to improve HIV care engagement — Based on the barriers to HIV care experienced by the pre-intervention cohort, we will design a system intervention to be implemented at the Radiotherapy Centre at Parirenyatwa Hospital. This intervention will include 2-3 components, each intended to improve engagement in HIV care or address specific barriers to HIV care. It may include strategies like improving documentation of HIV-related information in oncology patient records, improving processes for referrals and access to HIV-related prescriptions, and supporting better communication between oncology and HIV clinical care teams.
  Arms: Post-intervention cohort

SUMMARY:
In Zimbabwe, people who have cancer and HIV may have a difficult time staying engaged in their HIV care while they are being treated for cancer. This is because HIV and cancer care are usually provided at different health facilities, which can result in barriers to accessing clinical care for both HIV and cancer at the same time. It is important to remain engaged in HIV care, and continue taking medication to treat HIV throughout cancer treatment. The goal of this project is to identify barriers that make it difficult to stay engaged in HIV care and continue HIV treatment during cancer treatment and develop strategies to address them. The investigators will accomplish this by first observing a group of 150 people with cancer and HIV who are receiving cancer treatment at Parirenyatwa Hospital, in Harare, Zimbabwe. The investigators will measure barriers to accessing HIV care, and disruptions to HIV care engagement during cancer treatment. Next, the investigators will work with experts and key stakeholders to develop strategies that can be put in place at Parirenyatwa Hospital to better support engagement in HIV care during cancer treatment. The investigators will work with the cancer ward at the hospital to implement these strategies. Finally, the investigators will observe a second group of 150 people with cancer and HIV, who begin their cancer treatment at Parirenyatwa Hospital after the strategies have been put in place. The investigators will measure acceptability of these strategies to both patients and hospital staff. The investigators will also measure barriers to accessing HIV care and disruptions to HIV care engagement in the second group. The investigators will compare barriers to HIV care and HIV care engagement in the second group to the first group, to determine whether the strategies make it easier for people with cancer and HIV to remain engaged in HIV care during cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Registered patient at Parirenyatwa Hospital Radiotherapy Centre, receiving cancer treatment for a new diagnosis
* HIV-positive

Exclusion Criteria:

* Benign diagnosis or cancer recurrence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability of strategies to improve engagement in HIV care during cancer treatment | Acceptability assessed at Months 1, 3, and 6 after enrollment in pilot cohort
  Acceptability of the strategies to improve engagement in HIV care during cancer treatment will be assessed using questionnaires administered during 6 months of follow-up after enrollment in the post-intervention cohort. The primary outcome will only be assessed in the post-intervention cohort.

SECONDARY OUTCOMES:
Missed ART prescription refills | From enrollment through 6 months of follow-up or completion of cancer treatment
  We will measure missed ART prescription refills by self-reported ability to collect ART during cancer treatment
ART adherence | From enrollment through 6 months of follow-up or completion of cancer treatment
  We will measure ART adherence via self-reported missed ART doses, collected by questionnaire
Missed HIV clinical visits | From study enrollment through 6 months of follow-up or completion of cancer treatment
  We will measure missed HIV clinical visits by self-reported ability to attend HIV clinic visits during cancer treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michalina Montaño, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Parirenyatwa Hospital, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: No
This is not an individual intervention - the intervention under study will be to the health system